CLINICAL TRIAL: NCT02698592
Title: Comparative Study to Assess Safety and Efficacy of Catheters CelsiusTMDS® 8 mm, Thermocool® 3.5 mm of Irrigated Tip and Thermocool® SF in the Treatment of Cavo-tricuspid Isthmus Dependent Atrial Flutter
Brief Title: Evaluation of Thermocool SF Catheter on the Common Cavo-tricuspid Isthmus Dependent Atrial Flutter Ablation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Central de Asturias (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38/2012
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Atrial Flutter.
Keywords: atrial flutter; ablation; Thermocool SF catheter
MeSH Terms: conditions — Atrial Flutter | interventions — Catheters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CelsiusTMDS® 8 mm catheter (Active Comparator): 50 patients underwent ablation with CelsiusTMDS® 8 mm catheter.
  Interventions: Device: CelsiusTMDS® 8 mm catheter
- Thermocool® 3.5 mm irrigated catheter (Active Comparator): 50 patients underwent ablation with Thermocool® 3.5 mm catheter of irrigated tip.
  Interventions: Device: Thermocool® 3.5 mm catheter of irrigated tip
- Thermocool® SF catheter (Experimental): 50 patients underwent ablation with Thermocool® SF catheter.
  Interventions: Device: Thermocool® SF catheter

INTERVENTIONS:
Device: CelsiusTMDS® 8 mm catheter — After demonstrating cavo-tricuspidal isthmic dependant atrial flutter with a duodecapolar catheter, ablation with continuous tissue lesion will be performed with CelsiusTMDS® 8 mm catheter, until complete isthmic block is achieved.
  Arms: CelsiusTMDS® 8 mm catheter
Device: Thermocool® 3.5 mm catheter of irrigated tip — After demonstrating cavo-tricuspidal isthmic dependant atrial flutter with a duodecapolar catheter, ablation with continuous tissue lesion will be performed with Thermocool® 3.5 mm catheter of irrigated tip, until complete isthmic block is achieved.
  Arms: Thermocool® 3.5 mm irrigated catheter
Device: Thermocool® SF catheter — After demonstrating cavo-tricuspidal isthmic dependant atrial flutter with a duodecapolar catheter, ablation with continuous tissue lesion will be performed with Thermocool® SF catheter, until complete isthmic block is achieved.
  Arms: Thermocool® SF catheter

SUMMARY:
The purpose of this study is to determine whether the Thermocool SF ® system is at least as effective and safe as regular 8mm catheters and irrigated tip catheters in the treatment of cavo-tricuspid isthmus dependent atrial flutter.

DETAILED DESCRIPTION:
The catheter of Biosense Webster Thermocool SF® is characterized by a porous, thin-walled tip allowing a uniform cooling of the catheter tip and so, achieving increased efficiency in cooling. This allows to reduce the flow of irrigation and power output while achieving similar tissue temperatures as the conventional irrigated catheters. There is evidence of greater efficiency of Thermocool SF® catheter in causing tissue damage, but there are no clinical studies on the specific treatment of common atrial flutter.

Investigators hypothesize that the Thermocool SF® system is at least as effective and safe in the treatment of cavo-tricuspid isthmus dependent atrial flutter as conventional and 8 mm irrigated tip catheters.

150 patients with common atrial flutter were randomized to 3 groups of 50 patients and each group underwent ablation catheter ablation with CelsiusTMDS® 8 mm, 3.5 mm irrigated tip Thermocool® or Thermocool® SF respectively. After the procedure, patients are being followed by clinical reviews, electrocardiograms at the 3rd, 6th and 12th months, 24h ECG-Holter examination at the first and 6th month and monthly phone consultation. Rate of recurrence and presence of other supraventricular arrhythmias are being recorded during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic common atrial flutter.
* Electrocardiographic documentation of common atrial flutter.

Exclusion Criteria:

* Refusal to give consent.
* Life expectancy less than 6 months.
* Contraindication for ablation.
* Previous cavo-tricuspid isthmus ablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time to get cavo-tricuspid isthmus block | during the ablation.

SECONDARY OUTCOMES:
Time of fluoroscopy. | during the ablation.
Radio frequency application time. | during the ablation.
Complications. | within the first 24 hours.
  Defined as vascular complications, cardiac tamponade and outbursts by tissue boiling.
Recurrence of atrial flutter. | one year.

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Rubín López, PhD, Principal Investigator — Hospital Universitario Central de Asturias
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

REFERENCES:
- [Background] Tsai CF, Tai CT, Yu WC, Chen YJ, Hsieh MH, Chiang CE, Ding YA, Chang MS, Chen SA. Is 8-mm more effective than 4-mm tip electrode catheter for ablation of typical atrial flutter? Circulation. 1999 Aug 17;100(7):768-71. doi: 10.1161/01.cir.100.7.768. PMID 10449701
- [Background] Jais P, Shah DC, Haissaguerre M, Hocini M, Garrigue S, Le Metayer P, Clementy J. Prospective randomized comparison of irrigated-tip versus conventional-tip catheters for ablation of common flutter. Circulation. 2000 Feb 22;101(7):772-6. doi: 10.1161/01.cir.101.7.772. PMID 10683351
- [Background] Schreieck J, Zrenner B, Kumpmann J, Ndrepepa G, Schneider MA, Deisenhofer I, Schmitt C. Prospective randomized comparison of closed cooled-tip versus 8-mm-tip catheters for radiofrequency ablation of typical atrial flutter. J Cardiovasc Electrophysiol. 2002 Oct;13(10):980-5. doi: 10.1046/j.1540-8167.2002.00980.x. PMID 12435182
- [Background] Scavee C, Georger F, Jamart J, Mancini I, Collet B, Blommaert D, De Roy L. Is a cooled tip catheter the solution for the ablation of the cavotricuspid isthmus? Pacing Clin Electrophysiol. 2003 Jan;26(1P2):328-31. doi: 10.1046/j.1460-9592.2003.00043.x. PMID 12687839